CLINICAL TRIAL: NCT05499975
Title: Comprehensive Health Assessment for my Cancer Treatment Plan: Field Validation of a Geriatric Assessment Tool for Cancer Patients
Brief Title: Comprehensive Health Assessment for my Cancer Treatment Plan
Acronym: CHAMP-F
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 4011
Record Dates: First submitted 2022-08-02; First posted 2022-08-12 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Cancer; Older Adults
Keywords: geriatric assessment; older adults; cancer; treatment modification; supportive care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single-arm non-randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Older adults completing the CHAMP tool before treatment decision is made (Experimental): Eligible participants who consent to the study will be asked to complete questionnaires about socio-demographic characteristics, literacy, and technology comfort. Subsequently, participants will be asked to complete the CHAMP tool at home or in the clinic before their medical appointment with the oncologist. Next, participants will see their oncologist for their consultation. Approximately one week after the consultation, participants will be asked to complete 3 questionnaires about their experience and satisfaction with the CHAMP tool
  Interventions: Other: Self-reported online geriatric assessment (CHAMP)

INTERVENTIONS:
Other: Self-reported online geriatric assessment (CHAMP) — The CHAMP tool is a self reported online tool that has been developed to increase patients' accessibility to geriatric assessment and improve treatment decision making. The tool includes questions about function, mobility, cognition, nutrition, social support, depression substance use disorders, and miscellaneous items. Based on usability testing in the previous phase of this study, the tool can be completed in approximately 10-15 minutes. The tool generates a summary report with recommendations for patients and clinicians.

SUMMARY:
Geriatric assessment (GA) predicts treatment toxicity and overall mortality in older adults with cancer. To improve treatment decision making in older adults with cancer, the American Society of Clinical Oncology (ASCO) and the International Society of Geriatric Oncology recommend implementation of GA for all older adults with cancer. However, in-person GA may not be feasible in several institutions for various reasons, including lack of geriatricians and/or lack of time or resources. These challenges can be minimized through a self-reported online GA that can be completed by patients prior to their medical appointment. In a previous study, the investigators developed a self-reported online GA, known as the Comprehensive Health Assessment for My Cancer treatment Plan (CHAMP) that be used in geriatric oncology to increase accessibility to GA for older adults with cancer. In this study, our aim is to deploy the CHAMP tool to various oncology clinics across 4 institutions and assess feasibility outcomes, as well as the impact of the CHAMP tool on cancer treatment plan and supportive care strategies.

DETAILED DESCRIPTION:
Introduction:

Age, cancer, and under-treatment. Over 60% of cancer diagnoses and 71% of cancer deaths are in older adults (OAs) age 65+y. OAs are under-screened, under-diagnosed, under-staged, and under- treated for cancer compared to middle-aged individuals. Increasing age is associated with changing physiology along with increasing comorbidity, polypharmacy, functional impairment, and cognitive impairment. Frailty (reduced physiologic reserve) is common but not universal. The inability of oncologists to accurately 'stage the ageing' and separate frailty from healthy ageing leads to both over- treatment of many frail and under-treatment of many fit older adults around the world. To help clinicians and patients select appropriate cancer treatment(s) and identify issues that may affect treatment delivery, the American Society of Clinical Oncology and the Int'l Society of Geriatric Oncology (SIOG) recommend GA for OAs when cancer treatment is considered. A GA has 8 key assessment domains (i.e. comorbidity, functional status, medications, falls risk, nutrition, social supports, cognition, mood), each of which is relevant to cancer treatment.GA can change treatment decisions in almost 30% of patients, reducing over- and under-treatment, and allowing for personalization of cancer therapy. GA helps predict who is at high risk of treatment toxicity, enabling treatment modifications and/or additional supportive care, leading to reductions in severe toxicity of 10-20% and prolonged time on treatment. However, GA has not been widely implemented in oncology settings in most countries, in large part due to lack or limited availability of timely geriatric expertise. An attractive, scalable solution is a patient self-completed GA.

The investigators designed the CHAMP tool, a self-reported online GA that can be completed by older adults at home or in the clinic prior to their medical appointment. The process for developing CHAMP included the following steps: i) a systematic review and a Delphi Panel of expert clinicians to select the final domains and items/questionnaires; ii) design sessions with older adults with cancer to develop the layout and contact of the tool; iii) usability sessions with older adults with cancer to finalize the tool; and iv) design sessions with oncology clinicians to develop the tool's clinician interface. The CHAMP tool is now ready for field testing.

Our objectives are to measure feasibility outcomes and determine whether the CHAMP tool impact treatment decisions and supportive care strategies in older adults with cancer.

Methods:

A total of 210 older adults (65+y) with cancer of any type and stage will be recruited from 4 centres - 3 academic (Princess Margaret Cancer Centre, Odette Cancer Centre, St. Michael's) and 1 community site (St. Joseph's Health Centre). Older adults who agree to participate will be asked to provide information on sociodemographic characteristics and comfort with technology prior to completing the CHAMP tool. Subsequently, older adults will be asked to complete the tool either prior to clinic (at home via internet) or in clinic (via iPad) prior to their consultation with the oncologist. Following completion of the CHAMP tool and prior to recommending therapy, a member of the research team will provide the CHAMP results to the oncologist. The oncologist will be asked the proposed treatment plan and whether the patient is fit, vulnerable, or frail using standard definitions. Then, the oncologist will be asked of whether the treatment plan intent is being modified based on the CHAMP tool. The CHAMP tool also contains evidence-based recommendations for oncologists on strategies to reduce risk and address geriatric domains. Surveys will be used to assess patients' and oncologists' satisfaction with the tool.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 65 years and over referred to surgical oncology, radiation oncology, medical oncology at Princess Margaret Cancer Centre, St. Michael's Hospital, Sunnybrook Health Sciences, or St. Joseph's Health Centre.
2. Able to speak and understand English.
3. Able to provide informed consent.

Exclusion Criteria:

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 180 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Completeness of the CHAMP tool | Within one week from medical appointment
  Proportion of older adults who consented to the study who completed the CHAMP tool and had a discussion with their oncologist about the CHAMP results.
Time to fill out the CHAMP tool | Within one week from medical appointment
  In minutes, recorded via user interaction logs which will include data such as user's actions and interactions with the actual interface such as clicks, point-an-select actions, use of back button, etc.), and whether they completed it alone or needed help.
Satisfaction with the CHAMP tool | Older adults - within one week of their medical appointment. Oncologists - within one week of their last study patient.
  Measured via open-ended questions and a brief survey.

SECONDARY OUTCOMES:
Change in proposed treatment plan | Within 48 hours of their appointment with an older adults who has completed the CHAMP tool
  The impact of the CHAMP tool on proposed treatment plan will be measured through an adapted questionnaire which the investigators used in their previous studies. It measures if treatment was changed at all (yes/no), and if changed, then modified intensity, alternate modality, best supportive care only, or other.
Changes in supportive care strategies | Within 48 hours of their appointment with an older adult who completed the CHAMP tool
  The impact of the the CHAMP tool on supportive care strategies will be measured through a survey that will be completed by the treating oncologist. Additionally, the investigators will record the number of geriatric issues identified in the CHAMP summary and the number and type of recommendations provided to older adults and oncologists. The investigators will then review the charts of all older adults who completed CHAMP to abstract data on recommendations made by oncologists, referrals made to geriatrics and other health care providers, and other tests requested based on the recommendations.

CONTACTS AND LOCATIONS:
Overall Officials: Shabbir Alibhai, MD, Principal Investigator — University Health Network, Toronto; Martine Puts, PhD, Principal Investigator — University of Toronto
Locations (3):
- Canada (3):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Unity Health, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
The data of this study may be provided by the principal investigator upon reasonable request and upon approval of the IRB.